CLINICAL TRIAL: NCT03778502
Title: International Registry on the Use of the Direct Oral Anticoagulants for the Treatment of Unusual Site Venous Thromboembolism
Brief Title: DOAC in Unusual Site Venous Thrombosis
Acronym: DUST
Status: Completed | Type: Observational
Sponsor: University of Malta (Other)
Collaborators: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Nicoletta Riva, Lecturer, University of Malta
Other Study IDs: DUST
Record Dates: First submitted 2018-12-11; First posted 2018-12-19 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Splanchnic Vein Thrombosis; Cerebral Vein Thrombosis; Ovarian Vein Thrombosis; Renal Vein Thrombosis; Retinal Vein Thrombosis
MeSH Terms: conditions — Intracranial Thrombosis; Retinal Vein Occlusion | interventions — N(4)-oleylcytosine arabinoside; apixaban; Dabigatran; edoxaban; Rivaroxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Direct Oral Anticoagulants — Consecutive adult patients with objectively diagnosed unusual site venous thrombosis and treated with one of the DOAC (e.g. apixaban, dabigatran, edoxaban, rivaroxaban) will be eligible for this observational prospective registry
  Other Names: Apixaban; Dabigatran; Edoxaban; Rivaroxaban

SUMMARY:
Unusual site venous thromboembolism (VTE) refers to thrombosis occurring in venous districts outside the veins of the lower extremities and the pulmonary arteries, and includes splanchnic vein thrombosis (SVT), cerebral vein thrombosis (CVT), retinal vein thrombosis, ovarian vein thrombosis, and renal vein thrombosis. The use of the novel direct oral anticoagulants (DOAC), thrombin or factor Xa-inhibitors (such as dabigatran, apixaban, edoxaban, rivaroxaban), in patients with unusual VTE in clinical practice is increasing. Through an international multicentre prospective registry, the investigators aim to evaluate the rationale for the use of the DOAC for the treatment of unusual site VTE and to assess the safety and effectiveness of this approach in real life clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Objective diagnosis of venous thrombosis not involving the upper limbs, lower limbs and pulmonary arteries
* Treatment with one of the DOAC (e.g. apixaban, dabigatran, edoxaban, rivaroxaban)

Exclusion Criteria:

• Enrolment in interventional studies evaluating the DOAC for the treatment of unusual site VTE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients who fulfill the inclusion/exclusion criteria at the participating thrombosis centers will be eligible
Sampling Method: Non-Probability Sample
Enrollment: 358 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Rationale for the use of the direct oral anticoagulants | Baseline
  Possible reasons for choosing one of the direct oral anticoagulant (multiple choice question)

SECONDARY OUTCOMES:
Rate of major bleeding events | 12 months
Rate of vascular events | 12 months

CONTACTS AND LOCATIONS:
Locations (24):
- Henry Ford Health System, Detroit, Michigan, United States
- Ottawa Hospital Research Institute, Ottawa, Canada
- France (6):
  - CHU Amiens Picardie, Amiens
  - Hôpital de la Cavale Blanche, Brest
  - Hôpital Edouard Herriot, Lyon
  - Hopital Louis Mourier, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Centre Hospitalier Universitaire de Saint-Etienne, Saint-Etienne
- Sheba medical center, Tel Litwinsky, Israel
- Italy (9):
  - Azienda Ospedaliera Universitaria di Bologna, Bologna
  - Ospedale Maggiore, Bologna, Bologna
  - Ospedale Sant'Anna, ASST Lariana, Como
  - Ospedale Policlinico San Martino, Genova
  - Ospedale San Paolo, Milan
  - University Hospital of Padova, Padua
  - Catholic University, Rome
  - Sapienza Università di Roma, Rome
  - University of Insubria, Varese
- University of Malta, Msida, Malta
- Radboud University Medical Center Nijmegen, Nijmegen, Netherlands
- University Medical Centre Ljubljana, Ljubljana, Slovenia
- Spain (2):
  - Clinica Universidad de Navarra, Madrid
  - Virgen del Rocío Hospital and Instituto de Biomedicina, Seville
- King Chulalongkorn Memorial Hospital, Bangkok, Thailand